CLINICAL TRIAL: NCT02894996
Title: Does the Response to a Mini-fluid Challenge of 3ml/kg in 2 Minutes Predict Fluid Responsiveness for Elective Pediatric Anesthetized Patient?
Brief Title: Does the Response to a Mini-fluid Challenge of 3ml/kg in 2 Minutes Predict Fluid Responsiveness for Pediatric Patient?
Acronym: PEDIFLUID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL16_0444; 2016-A01192-49 (Other: ID-RCB)
Record Dates: First submitted 2016-09-04; First posted 2016-09-09 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Anesthesia
Keywords: pediatric; anesthesia; fluid responsiveness; hemodynamic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pediatric patient for general anesthesia (Other): Pediatric patients for general anesthesia elected for scheduled surgery Patients weight between 8 and 30 kilograms
  Interventions: Drug: fluid challenge

INTERVENTIONS:
Drug: fluid challenge — fluid challenge realized after induction of anesthesia at a steady state, to assess fluid responsiveness and correct hypovolemia. The usual fluid bolus of 15ml/kg in 10 minute will be fragmented in 2 fluid boluses (3ml/kg in 2 minutes followed by measurement of hemodynamic parameter after 1 minute of the end of the 1st fluid bolus and followed by 12 ml/kg in 8 minutes then followed by measurement of hemodynamic parameters after one minute after the end of the 2nd fluid fragmented fluid challenge. Total administered: 15 ml/kg in 11 minutes. end of the study at 12 minutes.
  Other Names: fluid bolus

SUMMARY:
To predict fluid responsiveness in anesthetized pediatric patient is not an easy task although anesthesia provider has to deal with this question on their daily practices. Today, very few parameters can help anesthesia provider to predict fluid responsiveness in the pediatric anesthetized patient. Therefore anesthesia provider are let with fluid challenge with high volume of fluid boluses to see if patient were fluid responsive or not. This could lead to fluid overload and it's associated morbidity. We would like to investigate if the cardiac output response to a mini fluid challenge of 3 ml/kg in 2 minutes would be predictive of the response to an usual fluid challenge of 15 ml/kg in 10 minutes in elective pediatric anesthetized patients.

DETAILED DESCRIPTION:
The main objective is to determine whether the new test "the stroke volume variation after fluid challenge of 3ml/Kg" provides information about fluid responsiveness namely increased cardiac output. This new test will be compared to "gold standard" that is, "the stroke volume variation after standard fluid challenge of 15ml/Kg". It is the evaluation of the diagnostic accuracy of a diagnostic test based on an index obtained by transthoracic cardiac echocardiography for diagnosing fluid responsiveness. This index is the stroke volume variation measured by transthoracic cardiac echography.

The study will include anesthetized patients undergoing scheduled surgery. For hemodynamic optimization, these patients will benefit, early after anaesthetic induction, before the surgical procedure has started, from a fluid challenge of 15ml/kg achieved in two stages (3 ml/Kg then 12 ml/kg) separated by an interval of one minute. Three-time hemodynamic will be analyzed.

* T0: basal
* T1: one minute after first vascular filling with 3ml/Kg in 2 minutes
* T2: one minute after second vascular filling with 12 ml/Kg in 8 minutes which is performed one minute after the end of the first filling (a total of 15 ml/kg)

At each time, we will retrieve a collection of hemodynamic data (stroke volume, cardiac output) obtained by transthoracic echocardiography, standard method to assess fluid responsiveness. And at the same times, the PVI and hemodynamic parameters obtained by esophageal Doppler will be noted.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patient for scheduled surgery
* from 8 to 30 kg of weight

Exclusion Criteria:

* denied from the child or their parents
* congenital cardiopathy
* cardiovascular shunt
* respiratory dysfunction
* hepatic dysfunction
* renal dysfunction
* intracranial hypertension

Ages: 6 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2018-02-02 (Actual); Study Completion 2018-02-02 (Actual)

PRIMARY OUTCOMES:
Stroke volume variation | 12 minutes
  The main objective is to determine whether the new test "the stroke volume variation after fluid challenge of 3mL/Kg" provides information about fluid responsiveness namely increased cardiac output. This new test will be compared to "gold standard" that is, "the stroke volume variation after standard fluid challenge of 15mL/Kg". It is evaluation of the diagnostic accuracy of a diagnostic test based on an index obtained by transthoracic echocardiography for diagnosing fluid responsiveness. This index is the stroke volume variation.

SECONDARY OUTCOMES:
Correlations between stroke volume variation after expansion of 3mL/Kg and after 15mL/Kg | 12 minutes
  To compare the correlations between stroke volume variation after volume expansion of 3 mL/kg and after volume expansion of 15 mL/kg
Diagnostic capacity of PVI and esophageal doppler | 12 minutes
  To assess the capacity of the PVI and of common parameters obtained by esophageal Doppler in diagnosing fluid responsiveness

CONTACTS AND LOCATIONS:
Overall Officials: Marc Lilot, MD, Principal Investigator — Hospices Civils de Lyon Direction de la Recherche Clinique et de l'Innovation
Locations (1):
- Hopital femme mere enfant, Bron, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zorio V, Lebreton T, Desgranges FP, Bochaton T, Desebbe O, Chassard D, Jacquet-Lagreze M, Lilot M. Does a two-minute mini-fluid challenge predict fluid responsiveness in pediatric patients under general anesthesia? Paediatr Anaesth. 2020 Feb;30(2):161-167. doi: 10.1111/pan.13793. Epub 2020 Jan 20. PMID 31858641